CLINICAL TRIAL: NCT07230262
Title: A Controlled Randomized Trial Comparing Multiport RObotic and Laparoscopic Surgery for Elective Colorectal Resections in IBD Patients
Brief Title: Trial Comparing Multiport RObotic and Laparoscopic Surgery for Elective Colorectal Resections in IBD Patients (ACRO-IBD)
Acronym: ACRO-IBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S70917 /B3222025001767/I/U
Record Dates: First submitted 2025-09-16; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: IBD - Inflammatory Bowel Disease
Keywords: Patients with inflammatory bowel disease (IBD); Colorectal surgery in IBD patients
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multiport RObotic surgery (Active Comparator): Surgical procedure performed using a robotic system.
  Interventions: Procedure: Robotic colorectal surgery
- laparoscopic surgery (Active Comparator): Surgical method that uses a slender camera inserted through small incisions,
  Interventions: Procedure: Laparoscopic colorectal surgery

INTERVENTIONS:
Procedure: Robotic colorectal surgery — Colorectal surgery using robotic procedure
  Arms: multiport RObotic surgery
Procedure: Laparoscopic colorectal surgery — Colorectal surgery using laparoscopic procedure
  Arms: laparoscopic surgery

SUMMARY:
The aim of this study is to better understand whether robotic surgery leads to better outcomes than laparoscopy in terms of complications, recovery and quality of life.

DETAILED DESCRIPTION:
This clinical trial compares two surgical techniques, robotic surgery and conventional laparoscopic surgery, for patients with inflammatory bowel disease (IBD) requiring elective colorectal surgery. Both approaches are minimally invasive and commonly used in clinical practice. This is a randomized trial: participants will be randomly assigned to one of the two techniques. A total of 110 patients will be enrolled.

This study will evaluate the role of robotic surgery in the surgical treatment of inflammatory bowel disease.

Three quality-of-life questionnaires will be completed: before the procedure and at 30 and 90 days post-procedure. Pain will also be assessed during the first three days post-procedure using a specific score called the VAS.

This study will be conducted exclusively at the University Hospitals Leuven.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. At least 18 years of age at the time of signing the Informed Consent Form (ICF)
3. Diagnosed with IBD and eligible for elective minimally invasive colorectal surgery, including:

   1.4 Ileocecal/ileocolic resections 1.5 Segmental colectomies 1.6 Total colectomy 1.7 Proctocolectomy 1.8 Proctectomy
4. Procedures involving primary anastomosis or temporary or permanent stoma creation
5. Suitable for minimally invasive surgery

Exclusion Criteria:

1. Non IBD patients
2. Urgent surgery (<24 hours from hospital admission)
3. Not suitable for minimally invasive surgery
4. Ileoanal pouch construction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative morbidity | During the first 90 days postoperatively
  Assessed using the Comprehensive Complication Index (CCI)

SECONDARY OUTCOMES:
Conversion to open surgery | Surgery day
  Robotic/laparoscopic surgery to open surgery
2. Postoperative pain | First three postoperative days
  Pain measured according to the visual analogue scale (VAS). The minimum score is 0, the maximum score is 10. The lower the score (e.g. 1 or 2) the less pain; the higher the score (e.g. more than 7) the more pain.
Quality of life (QoL) | At 30 and 90 days postoperatively
  QoL using the SF-36 Physical Health Component
Costs | Till 90 days postoperatively
  Direct Medical Costs (Hospital-Based) & Indirect Hospital Costs

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Bislenghi, Professor, Principal Investigator — UZ Leuven
Locations (1):
- Abdominal Surgery, Leuven, Vlaams Brabant, Belgium